CLINICAL TRIAL: NCT00586261
Title: Does Chronic Thiazolidinedione Therapy Improve Endothelial Function and Preserve Renal Function in Non-Diabetic Patients With Chronic Kidney Disease?
Brief Title: Does Thiazolidinedione Therapy Improve Endothelial Function and Preserve Renal Function
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment because of the specifics of the inclusion criteria
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Patricia J M Best, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 06-002245
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Results first posted 2013-03-07 (Estimated); Last update posted 2013-03-15 (Estimated); Status verified 2013-03

CONDITIONS: Chronic Kidney Disease
Keywords: Kidney Failure, Chronic; Renal Insufficiency, Chronic; Proteinuria; Albuminuria
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic; Proteinuria; Albuminuria | interventions — Pioglitazone; Nitroglycerin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo 30 mg daily for 6 months, nitroglycerin was given to check the brachial reactivity.
  Interventions: Drug: Placebo; Drug: Nitroglycerin
- Pioglitazone (Active Comparator): Pioglitazone 30 mg daily for 6 months, nitroglycerin was given to check the brachial reactivity.
  Interventions: Drug: Pioglitazone; Drug: Nitroglycerin

INTERVENTIONS:
Drug: Pioglitazone — Pioglitazone 30 mg daily for 6 months
  Other Names: Actos
  Arms: Pioglitazone
Drug: Placebo — Placebo 30 mg daily for 6 months
  Arms: Placebo
Drug: Nitroglycerin — 0.4 mg sublingual nitroglycerin tablet was given to all patients without a contraindication to check the brachial reactivity.
  Other Names: Nitrostat

SUMMARY:
The hypothesis of the current proposal is that chronic pioglitazone therapy will result in improved endothelial function, decreased inflammation, and preservation of renal function in patients with CKD but without diabetes.

DETAILED DESCRIPTION:
Despite continued improvements in the outcomes of patients with cardiovascular disease, similar improvements have not been seen in patients with chronic kidney disease (CKD). CKD constitutes one of the highest risk populations for cardiovascular disease. When the creatinine clearance is ≤ 60 ml/min the risk for cardiovascular events is greater than that of diabetes. However, few studies have focused on the prevention or treatment of coronary artery disease (CAD) in CKD patients.

The development of endothelial dysfunction and increased inflammation appear to be critical in the development of atherosclerosis and cardiovascular disease. The broad long-term objective of this grant proposal is to determine unique therapies to reduce endothelial dysfunction and inflammation, and thereby help to prevent cardiovascular disease and preserve renal function in patients with CKD. Thiazolidinediones such as pioglitazone appear to improve endothelial function and decrease inflammation, an effect that may be present in patients with or without diabetes.

To address this hypothesis the following Specific Aims are proposed:

1. To determine the effects of chronic pioglitazone therapy on endothelial function in non-diabetic patients with CKD (creatinine clearance ≤ 60 ml/ min, but not on dialysis)
2. To determine the effects chronic pioglitazone therapy on inflammation and oxidative stress in non-diabetic patients with CKD
3. To determine the effects chronic pioglitazone therapy on progression of renal disease in non-diabetic patients with CKD

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years.
* Creatinine clearance ≤ 60 ml/min by the Cockcroft-Gault equation
* Patients not anticipated to go on dialysis or have renal transplantation in the next 6 months
* Ability to provide informed consent
* Life expectancy greater than 12 months

Exclusion Criteria:

* Diabetes mellitus or a fasting blood glucose ≥ 110 mg/dL
* Acute renal failure
* Class 3 or 4 heart failure
* Liver failure, ascites, or an aspartate aminotransferase (AST) or alanine aminotransferase (ALT) two times the upper limit of normal
* Hemoglobin less than 9 mg/dL
* Multiple myeloma
* Premenopausal women not using at least 1 form of birth control
* Pregnant or nursing women
* Prisoners
* Known allergy to pioglitazone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2006-03; Primary Completion 2009-01 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia M. Best, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the Mayo Clinic, Rochester, Minnesota.
Period: Overall Study
Arm/Group | Pioglitazone | Placebo
Started | 17 | 19
Completed | 17 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Pioglitazone Arm: study the specific dose of pioglitazone 30 mg daily for 6 months
  pioglitazone : pioglitazone 30 mg daily for 6 months
- Placebo Arm: study the specific dose of placebo 30 mg daily for 6 months
  placebo : placebo 30 mg daily for 6 months
- Total: Total of all reporting groups
Arm/Group | Pioglitazone Arm | Placebo Arm | Total
Number analyzed (Participants) | 17 | 19 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 4 | 7
  >=65 years | 14 | 15 | 29
Age Continuous [Mean (Standard Deviation); unit: years] | 74.2 (7.4) | 72.1 (8.3) | 73.1 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 10 | 10 | 20
Region of Enrollment [Number; unit: participants]
  United States | 17 | 19 | 36

OUTCOME MEASURES:

1. Primary Outcome: Change in Brachial Arterial Reactivity
Description: Brachial arterial reactivity was measured by ultrasound. A blood pressure cuff was placed around the right forearm. Using the ultrasound probe of the ultrasound, 2-dimensional images clearly defining the anterior and posterior intimal wall of the brachial artery were collected. Flow velocities were then measured using pulsed wave Doppler. The blood pressure cuff previously placed around the patient's right forearm was inflated to 200 mmHg. The cuff remained inflated for 5 minutes as the patient remained motionless and quiet. Prior to deflation, the patient was asked to remain still as flow velocities and 2-dimensional images were obtained immediately following cuff deflation. Then a 0.4 mg sublingual nitroglycerin tablet was given to all patients without a contraindication and all measurements were repeated.
Time Frame: After 6 months of treatment
Population: The study was stopped early due to low recruitment and no evidence of an effect in this analysis.
Measure: Mean (Standard Error); unit: mm
Arm/Group | Pioglitazone Arm | Placebo Arm
Number analyzed (Participants) | 17 | 19
mm | 0.8476 (1.35) | 2.6058 (1.35)

ADVERSE EVENTS:
Groups:
- Pioglitazone: Pioglitazone 30 mg daily for six months
- Placebo: Placebo 30 mg daily for six months
Arm/Group | Pioglitazone | Placebo
Serious Adverse Events (participants affected / at risk) | 1/17 | 0/19
Other Adverse Events (participants affected / at risk) | 1/17 | 0/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pioglitazone (N=17) | Placebo (N=19)
hypoglycemia (Endocrine disorders) | 1 (1) | 0 (0) — One patient got low blood glucoses and discontinued the medication
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pioglitazone (N=17) | Placebo (N=19)
edema (Vascular disorders) | 1 (1) | 0 (0) — One patient got edema resulting in discontinuation.

LIMITATIONS AND CAVEATS:
The study was stopped early due to low enrollment because of the specifics of the inclusion criteria.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No